CLINICAL TRIAL: NCT06023069
Title: Preoperative Walking Evaluation and Postoperative Outcome in Non-cardiac Surgery
Brief Title: Preoperative Walking Evaluation and Postoperative Outcome
Acronym: PREVENT
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Max Bell, MD, PhD, Karolinska Institutet
Other Study IDs: N32276 PMI/Karolinska
Record Dates: First submitted 2023-08-28; First posted 2023-09-05 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: General Surgery; Perioperative Medicine
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Number of steps recorded by mobile phone as a proxy for physical activity — This cohort is likely to have patients with many steps/day (high activity) and few steps/day (low activity)

SUMMARY:
The hypothesis is that physical activity is associated with a reduced risk of complications and death after surgery.

Self-reporting of physical activity is prone to be unreliable. In order to obtain a better picture of patients' physical activity, we intend to investigate the association between the average number of steps and postoperative outcomes. Many other objective measures of physical activity are costly and time-consuming to perform; for example, exercise tests, extensive sampling, and longer questionnaires.

The primary research question is: Do patients with a higher degree of physical activity, measured as the average number of steps recorded on the patient's mobile phone, have a reduced risk of peri/postoperative complications and death, measured as Days At Home alive at 30 days (DAH30)?

Secondary research questions include:

Is physical activity, measured as the average number of steps recorded on the patient's mobile phone, linearly linked to DAH30? Is physical activity, measured as the average number of steps recorded on the patient's mobile phone, associated with specific peri/postoperative organ impact, such as lung, heart, cerebral, infection, or kidney complications? Is physical activity, measured as the average number of steps recorded on the patient's mobile phone, also linked to long-term outcomes one year after surgery? Is physical activity, measured as the average number of steps recorded on the patient's mobile phone, solely associated with DAH30 and organ complications for specific patient groups in terms of age, comorbidities, and/or type of surgery?

DETAILED DESCRIPTION:
Project Description Method This is a non-interventional prospective observational multicenter study of the association between physical activity and peri/postoperative outcomes, planned to be conducted in two stages. First, as a pilot study involving multiple participating anesthesia/surgery clinics. Following this, the plan is to analyze data from the mentioned pilot study and then launch a global multicenter study on a more defined patient group.

Procedures/Data Collection Preoperatively: The investigators will record age, gender, comorbidities, and ongoing medication, as well as ASA classification, frailty score, and mDASI (modified Duke Activity Status Index), which is a measure of functional ability. Routine preoperative laboratory tests will be noted. Furthermore, the investigators intend to record average physical activity, including daily step count on average at one, six, and twelve months before surgery, based on data from the patient's mobile phone*. Type of planned surgery will be recorded.

*The dominant mobile phones on the market (iOS and Android-based) use different types of systems to count steps. Some mobile phones completely lack such systems. The validation of how accurately they count steps per day also varies. We will record the model and operating system, as well as the type of app used. Not all patients carry their phones all the time; we intend to register their own estimate of how often it is carried. A few patients do not have a mobile phone and cannot contribute step per day data.

Intraoperatively: The investigators will record anesthesia method, operation time (incision time and total operation time), fluid balance, bleeding, and transfusion requirements, as well as adverse events such as blood pressure drops, hypoxia, tachycardia.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (equal to or over 18 years) undergoing elective non-cardiac surgery providing informed consent

Exclusion Criteria:

Patients that can not provide informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients (equal to or over 18 years) undergoing elective non-cardiac surgery
Sampling Method: Probability Sample
Enrollment: 264 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
DAH30 (Days At Home alive at 30 days) | 30 days after index surgery
  DAH30: Patients who are hospitalized for 14 days postoperatively but are alive on day 30 will have DAH30=16. Patients who are hospitalized for five days, then discharged, but return after 10 days for an additional 11-day stay, will have DAH30=14. Anyone who dies within 30 days will have DAH30=0. This outcome measure is validated in several studies and has a significant advantage in that it correlates well with complications, even better than length of stay (LOS)

SECONDARY OUTCOMES:
Mortality | Mortality will be recorded at 30, 60, 90 and 365 days after index surgery
  Death within the time frames described below

CONTACTS AND LOCATIONS:
Overall Officials: Max Bell, Principal Investigator — N32276 PMI/Karolinska
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided